CLINICAL TRIAL: NCT01984671
Title: Home-Based Tablet Computer Pain Coping Skills Following Stem Cell Transplant
Brief Title: mPCST for BMT Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00047952
Record Dates: First submitted 2013-10-31; First posted 2013-11-15 (Estimated); Results first posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Stem Cell Transplant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile pain coping skills training (mPCST) (Experimental): Participants in this condition completed the first session following their baseline survey assessment. The developed mPCST protocol included 1 in-person session at the medical center between the patient and study therapist, which led to the development of a successful working relationship and the integration of mPCST with the patient's medical care. Then, once the patient returned home following intensive outpatient care, 5 more sessions were conducted using videoconferencing. Last, participants completed the post-assessment.
  Interventions: Behavioral: Mobile Pain Coping Skills Training
- Usual care control (No Intervention): Patients in this condition will have access to activity tracker syncing and daily symptoms assessment following their baseline survey assessment. HCT education participants will be encouraged to download the Transplant (HCT) Guidelines mobile app that is free of charge. Last, participants completed the post-assessment.

INTERVENTIONS:
Behavioral: Mobile Pain Coping Skills Training
  Arms: Mobile pain coping skills training (mPCST)

SUMMARY:
We used a small randomized controlled trial (n=36) to compare a Mobile Health Pain Coping Skills (mPCST) to Usual Treatment for patients having received hematopoietic stem cell transplant.

DETAILED DESCRIPTION:
The investigator proposes to develop and test a Mobile Health Pain Coping Skills (mPCST) protocol for HSCT patients with persistent pain to meet the challenges of HSCT patients with pain as they transition from hospital based care to their home environment. We used a small randomized controlled trial to examine the feasibility and acceptability, and engagement in the developed mPCST protocol. We compared the effects of usual care to the developed mPCST protocol on pain disability, pain self-efficacy, fatigue, and physical disability.

ELIGIBILITY:
Inclusion Criteria:

1. receipt of an stem cell transplant due to an oncological disease,
2. no prior stem cell transplant,
3. report a clinical pain score of at least 3/10, and
4. an age of > 21.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-10-02 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Somers TJ, Kelleher SA, Dorfman CS, Shelby RA, Fisher HM, Rowe Nichols K, Sullivan KM, Chao NJ, Samsa GP, Abernethy AP, Keefe FJ. An mHealth Pain Coping Skills Training Intervention for Hematopoietic Stem Cell Transplantation Patients: Development and Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 Mar 19;6(3):e66. doi: 10.2196/mhealth.8565. PMID 29555620

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mobile Pain Coping Skills Training (mPCST) | Usual Care Control
Started | 18 | 18
Completed | 16 | 17
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Pain Coping Skills Training (mPCST) | Usual Care Control | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Full Range); unit: years] | 54.6 [29 to 70] | 57.9 [40 to 75] | 56.25 [29 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 7 | 11 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Measured by the Overall Percentage of Completed Sessions
Description: Presented as the (total number of completed sessions for all participants) divided by the (total number of planned sessions for all participants) multiplied by 100. The goal of this study was to develop a PCST intervention that could be used to enhance the ability of HCT patients to manage their pain following transplant, that is feasible and acceptable.
Time Frame: 10 weeks
Population: Usual care participants did not attend sessions.
Measure: Number; unit: percentage of sessions
Units Other Than Participants: mPCST sessions
Arm/Group | Mobile Pain Coping Skills Training (mPCST) | Usual Care Control
Number analyzed (Participants) | 18 | 0
Number analyzed (mPCST sessions) | 108 | 0
percentage of sessions | 83 |

2. Secondary Outcome: Cohen's D Effect Size of the Change in Pain Disability From Baseline to 10 Weeks
Description: A positive value indicates improvement in pain disability and a negative value indicates a decline.
Time Frame: Baseline to 10 weeks
Measure: Number; unit: Cohen's d
Arm/Group | Mobile Pain Coping Skills Training (mPCST) | Usual Care Control
Number analyzed (Participants) | 18 | 18
Cohen's d | 0.79 | 0.69

3. Primary Outcome: Acceptability as Measured by the Percentage of Participants Who Responded in the Affirmative for Each Item on the Assessment
Description: The goal of this study was to develop a PCST intervention that could be used to enhance the ability of HCT patients to manage their pain following transplant, that is feasible and acceptable.
Time Frame: 10 weeks
Population: Usual care participants did not attend sessions.
Measure: Number; unit: percentage of participants
Arm/Group | Mobile Pain Coping Skills Training (mPCST) | Usual Care Control
Number analyzed (Participants) | 18 | 0
percentage of participants
  Helpful (reported in assessment) | 80 |
  Easy to understand (reported in assessment) | 100 |
  Acceptable (reported in assessment) | 100 |

4. Secondary Outcome: Cohen's D Effect Size of the Change in Pain Self-efficacy From Baseline to 10 Weeks
Description: A positive value indicates improvement in pain self-efficacy and a negative value indicates a decline.
Time Frame: Baseline to 10 weeks
Measure: Number; unit: Cohen's d
Arm/Group | Mobile Pain Coping Skills Training (mPCST) | Usual Care Control
Number analyzed (Participants) | 18 | 18
Cohen's d | 0.61 | 0.10

5. Secondary Outcome: Cohen's D Effect Size of the Change in Fatigue From Baseline to 10 Weeks
Description: A positive value indicates improvement in pain self-efficacy and a negative value indicates a decline.
Time Frame: Baseline to 10 weeks
Measure: Number; unit: Cohen's d
Arm/Group | Mobile Pain Coping Skills Training (mPCST) | Usual Care Control
Number analyzed (Participants) | 18 | 18
Cohen's d | 0.94 | 0.81

6. Secondary Outcome: Cohen's D Effect Size of the Change in 2-minute Walk Test From Baseline to 10 Weeks
Description: A positive value indicates improvement in the 2-minute walk test and a negative value indicates a decline.
Time Frame: Baseline to 10 weeks
Measure: Number; unit: Cohen's d
Arm/Group | Mobile Pain Coping Skills Training (mPCST) | Usual Care Control
Number analyzed (Participants) | 18 | 18
Cohen's d | 0.66 | 0.41

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Mobile Pain Coping Skills Training (mPCST) | Usual Care Control
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No